CLINICAL TRIAL: NCT06279559
Title: Evaluating the Impact of Music Therapy on Psychological Well-being During High-risk Pregnancy
Brief Title: Music Therapy and High-risk Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Cristina Venturino, Dr, Istituto Giannina Gaslini
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTinHRP_v1_10/01/2023
Record Dates: First submitted 2024-02-14; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: High Risk Pregnancy
Keywords: music-therapy; high-risk pregnancy; attachment bond
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clinical experimental group (Experimental): pregnant women with the risk of preterm birth who will undergo music therapy intervention
  Interventions: Behavioral: Music-therapy
- clinical control group and non-clinical control group (No Intervention): pregnant women with the risk of preterm birth who will receive the usual ward care and pregnant women with pregnancy with a physiological course

INTERVENTIONS:
Behavioral: Music-therapy — 10 sessions of online music therapy held by expert music therapists
  Arms: clinical experimental group

SUMMARY:
The objective of this clinical trial is to assess the impact of a music therapy intervention on reactive psychological components related to the risk of preterm birth in hospitalized pregnant women. The primary inquiries it seeks to address are:

1. Can a music therapy intervention during high-risk pregnancy mitigate reactive psychological components (perceived emotional state, state anxiety and trait anxiety, depressive symptoms, perceived stress) related to the risk of preterm birth in hospitalized pregnant women?
2. Does music therapy intervention during high-risk pregnancy positively influence the development of the attachment bond between the mother and the child?
3. How does the risk of preterm birth modulate the future attachment bond between mother and child?

Participants will be categorized into three groups: a clinical experimental group (pregnant women at risk of preterm birth undergoing music therapy intervention), a clinical control group (pregnant women at risk of preterm birth receiving standard ward care), and a non-clinical control group (pregnant women with a physiologically progressing pregnancy).

Upon signing the informed consent, all three groups will be required to complete five self-report questionnaires assessing perceived positive and negative feelings, depressive symptoms, state anxiety and trait anxiety, perceived stress, and the mother-fetus attachment bond. Subsequently, the clinical experimental group will undergo ten online music therapy sessions, while the clinical control group will receive routine ward care. Following the music therapy sessions, both clinical groups will reassess the aforementioned measures. The non-clinical control group will complete the same self-report questionnaires with the same timing as the clinical groups. All three groups will be contacted three months after childbirth to complete a self-report questionnaire evaluating the postnatal attachment bond.

Researchers will compare the outcomes of the two clinical groups to address the first two research questions, while the comparison between the clinical control group and the non-clinical control group outcomes will be employed to answer the third research question.

DETAILED DESCRIPTION:
Background and Rationale Every year, approximately 15 million children are born prematurely worldwide, with a global incidence of around 11%. Preterm birth occurs when labor takes place between the 22nd and 37th completed weeks of gestation, representing a significant public health concern. Preterm birth is associated with higher rates of infant morbidity and mortality, increased risk of long-term medical complications, impaired neurological development, family stress, and substantial social costs. Conversely, the risk of preterm birth is a stressful event for caregivers, particularly for pregnant women, potentially evolving into a traumatic experience, eliciting feelings of anxiety and depression. In cases of preterm birth risk, the initial phase of parenthood is marked by uncertainty, dominated by prevalent emotional correlates of anxiety and fear of death, which, in turn, diminish the psychological investment in the child. Many parents respond to this reality with an initial phase of rejection and ambivalence towards the child, expressing both frustration and common concerns about the infant's survival.

The risk of preterm birth falls under high-risk pregnancies, defined as "[...] any unexpected or unforeseen medical or obstetric condition associated with pregnancy with an actual or potential risk to the health or well-being of the mother or fetus...". Compared to women with low-risk pregnancies, those with high-risk pregnancies exhibit significantly higher levels of stress and anxiety, report more negative emotions when facing stress, and have a worse emotional state. Additionally, women confined due to high-risk pregnancies show predominant emotional responses of fear, anxiety, and emotional distance from the child, along with depressive symptoms and feelings of loneliness. Thus, the emotional impact of the risk of preterm birth on pregnant women demands adequate clinical attention, particularly considering that the reactive symptoms mentioned above serve as predictive factors when exploring the psychosocial determinants of preterm birth.

Furthermore, the risk of preterm birth can negatively influence the development of the mother-fetus attachment bond (or prenatal attachment), although some studies report contrasting results. Prenatal attachment, derived from John Bowlby's Attachment Theory, is defined as "the emotional bond that normally develops between the pregnant parent and their unborn child". It serves as an early indicator of the future quality of the mother-child attachment bond and is a crucial factor influencing the child's subsequent well-being. Women with high-risk pregnancies may experience guilt for their condition, and the risk of preterm birth and premature rupture of membranes can interrupt the psychological preparation process for motherhood. Negative thoughts in pregnant women related to fetal health and the possibility of fetal death can evoke fear of developing a relationship with the fetus, hindering attachment development.

Therefore, it becomes crucial to identify effective, non-invasive, and adaptable methods within the hospital setting to reduce unpleasant emotional states in pregnant women at risk of preterm birth and promote the structuring of the attachment bond. In this context, recent research has increasingly focused on music therapy as one of the potential approaches to alleviate emotional states linked to pregnancy.

The World Federation of Music Therapy defines music therapy as "[...] the professional use of music and its elements as an intervention in medical, educational, and social environments with individuals, groups, families, or communities seeking to optimize their quality of life and improve physical, social, communicative, emotional, intellectual, and spiritual health". Recent literature reviews and meta-analytical studies have documented how music therapy can be effective in reducing stress-related symptoms (both in medical and mental health contexts), decreasing depressive symptoms, and anxious symptoms. Regarding its use during pregnancy, music therapy, besides significantly reducing mental health problems such as anxiety, depressive symptoms, and perceived stress in pregnant women, can address the sensory, physical, and emotional needs of pregnant women and support the process of creating the attachment bond, promoting the development of meaningful interactions.

In conclusion, the risk of preterm birth requires prolonged hospitalization for pregnant women. It can have a high impact on both individual and couple's emotional and psychological well-being, as well as on the construction of the mother-child relationship. Hospitalization, while serving as a protective element and monitoring for the health of the unborn, intensifies fears and anxieties, inducing a "medicalization" that may be accompanied by feelings of inadequacy and helplessness. This, coupled with concerns about the effects of gestational complications on the fetus, can negatively influence the adaptation process to pregnancy and the development of the mother-child attachment. However, although numerous studies have delved into the topic of prenatal mother-child attachment development in normal pregnancies, the development of this relationship in high-risk pregnancies remains understudied. Additionally, to the best of our knowledge, the potential benefit of music therapy on the mental health of women with high-risk pregnancies and on pre- and post-natal attachment bonding is still underexplored in the literature of the field.

STUDY OBJECTIVES - Primary Objectives: The primary aim is to evaluate the effect of a music therapy intervention on reactive psychological components associated with the risk of preterm birth in hospitalized pregnant women.

The key psychological components of interest in this study include depressive symptoms, anxious symptoms, perceived stress, perceived well-being, prenatal attachment, and postnatal attachment.

- Secondary Objectives:

The secondary objectives are as follows:

1. - Assessment of Attachment Quality: To assess whether there are variations in the quality of pre-and postnatal attachment in hospitalized pregnant women at risk of preterm birth who do not undergo music therapy compared to pregnant women with uncomplicated pregnancies.
2. - Psychosocial Well-being: To identify aspects of psychosocial well-being influenced by music therapy intervention and those that do not appear to be affected.
3. - Timing of Intervention: To investigate whether differences in the gestational age at which music therapy intervention is conducted play a significant role in treatment efficacy.
4. - Pregnancy Characteristics and Personal History: To explore whether different aspects of the current pregnancy and the pregnant woman's personal, pathological, and physiological history, encompassing both behavioural and emotional factors, influence the effectiveness of the treatment.
5. - Demographic Variables: To examine whether sociodemographic variables influence the outcomes of music therapy intervention.

STUDY SETTING AND EXPERIMENTAL PHASES

Setting and Participant Recruitment:

To assess the effectiveness of the music therapy intervention, all consecutively hospitalized patients with a high risk of preterm birth at the Obstetrics and Gynecology Unit of I.R.C.C.S. Giannina Gaslini will be enrolled. They will be randomly assigned to either the experimental or control group. Additionally, to examine the impact of the preterm birth risk on the formation of attachment bonds, pregnant women with uncomplicated pregnancies attending check-ups at the same unit will be consecutively recruited. The sample will be recruited based on predefined inclusion criteria. Once invited to participate and after obtaining consent, patients will be recruited for the study.

Administration and Recruitment Phases:

The test administration phases will take place in the inpatient rooms of the Obstetrics and Gynecology Unit, in a protected setting, and/or through telecommunication methods. Music therapy interventions will be conducted exclusively via telecommunication.

1. st Phase: Patients will be asked for authorization to participate in the study. A detailed explanation of the study procedures, structured and identical across participants, will be provided to avoid influencing test completion or participant behaviour. The experimenter will ask patients to read and sign the study information sheet, informed consent form, and data processing consent. A patient will be considered enrolled only after obtaining authorization.
2. nd Phase: In the second phase, all participants will be asked to complete a form for collecting demographic and medical data along with six self-report questionnaires assessing perceived subjective well-being (PANAS), characteristics of mother-fetus attachment or prenatal attachment (MAAS), perceived stress levels (PSS), mood deflection and depressive symptoms (EPDS), and state and trait anxiety components (STAI-Y).
3. rd Phase: The third phase involves the music therapy intervention, exclusively for participants assigned to the clinical experimental group. Specifically, participants in the clinical experimental group will undergo a series of 10 music therapy sessions conducted by Dr. Francesca Pasini and Dr. Alessandra Ravizza. These sessions will be conducted via telecommunication and will have a high degree of structure in terms of both the course and content. Conversely, all other participants will receive standard ward care.
4. th Phase: Within one week after the conclusion of the music therapy intervention (to which only the experimental clinical group will be subjected), all participants will be asked to complete the self-report questionnaires administered during the 2nd phase again.
5. th Phase: All the participants will be contacted via email for a follow-up to assess the characteristics of mother-infant attachment or postnatal attachment (MPAS) three months after childbirth.

Timeline:

The duration of the two data collection sessions (pre and post-treatment) will mirror that of the standard session (approximately 50 minutes) as measurements will be taken during clinical hours. Each music therapy session will last approximately 75 minutes. It is noteworthy that the number of music therapy sessions will depend on the patient's therapeutic progress, availability, and treatment timing at the enrollment date.

ELIGIBILITY:
Inclusion Criteria (clinical groups):

* Age over 18 years old
* Adequate knowledge of the Italian language
* Consent to participate
* Condition of risk of preterm birth

Exclusion Criteria (clinical groups):

* Positive history of mental retardation
* Difficulty understanding the Italian language
* Presence of diagnosis of psychiatric pathology
* Absence of informed consent

Inclusion Criteria (non-clinical group):

* Age over 18 years old
* Adequate knowledge of the Italian language
* Consent to participate

Exclusion Criteria (non-clinical group):

* Positive history of mental retardation
* Difficulty understanding the Italian language
* Presence of diagnosis of psychiatric pathology
* Absence of informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | administered before and within one week after the conclusion of the music therapy intervention
  Edimburg Prenatal Depression Scale (EPDS)
State anxiety and trait anxiety | administered before and within one week after the conclusion of the music therapy intervention
  State-Trait Anxiety Inventory - Forma Y (STAI-Y)
Perceived stress | administered before and within one week after the conclusion of the music therapy intervention
  Perceived Stress Scale (PSS)
Perceived positive and negative feelings | administered before and within one week after the conclusion of the music therapy intervention
  Positive and Negative affect Schedule (PANAS)
Mother-fetus attachment bond | administered before and within one week after the conclusion of the music therapy intervention
  Maternal Antenatal Attachment Scale (MAAS)
Mother-child attachment bond | administered three months after the childbirth
  Postpartum Attachment Scale (MPAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Giannina Gaslini, Genova, Italy